CLINICAL TRIAL: NCT00551850
Title: A Phase I, Multi-Center, Dose-Escalation Trial to Determine the Safety, Tolerability, and Maximum Tolerated Dose of AV-412 Administered Orally Three Times Weekly to Subjects With Advanced Solid Tumors
Brief Title: A Safety Study of an Oral EGFR Inhibitor, AV-412, Administered Three Times Weekly in Advanced Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-412-07-102
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Cancer; Refractory Cancer
Keywords: epidermal growth factor inhibitor; solid tumors; advanced cancer
MeSH Terms: conditions — Neoplasms | interventions — MP 412

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AV-412

INTERVENTIONS:
Drug: AV-412 — oral solid dosage form administered three times weekly for 4 weeks (1 cycle)

SUMMARY:
The Epidermal Growth Factor Receptor (EGFR) is a validated target for the treatment of cancer, and agents targeting EGFR such as erlotinib (Tarceva®) are approved by the FDA for treatment of various solid tumors. AV-412 is a novel inhibitor of the EGFR-tyrosine kinase, with added activity against Her2 and other oncogenic kinases. Based on evidence of preclinical activity in various solid tumors, AV-412 is being developed as a possible novel treatment for cancer in humans.

PURPOSE: The purpose of this study is to test the safety and tolerability of AV-412, and determine the maximum tolerated dose of AV-412 when administered orally three times weekly.

DETAILED DESCRIPTION:
This is an open-label, dose escalation trial, and all subjects will receive oral AV-412 administered three times weekly or once weekly for 4 weeks (1 cycle) to evaluate safety and tolerability of AV-412. Treatment duration will be a minimum of 2 consecutive dosing cycles (8 weeks), if tolerated.

* Upon completion of the 2 cycles, subjects with documented stable disease or an objective response may continue to receive therapy at the same dose and schedule previously utilized, as long as tolerability is acceptable, for up to 1 year. Treatment beyond 1 year from the time of enrollment will be reviewed on a case-by-case basis between the sponsor and investigator.
* Subjects experiencing unacceptable toxicities or with documented disease progression will be discontinued from further participation in the study Accrual to next cohort will occur only after acceptable tolerance has been demonstrated throughout Cycle 1, and only after consultation with medical monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give written informed consent
2. 18 years and older
3. Evaluable disease or measurable disease according to RECIST.
4. Subjects enrolled in the MTD Cohort B must have the following:

   * A diagnosis of non-small cell lung carcinoma (NSCLC)
   * Received prior therapy with erlotinib or gefitinib for a minimum of 12 weeks
   * Demonstrated disease stabilization or an objective response during that prior treatment
   * Evidence of disease progression and measurable disease, according to RECIST
5. Histologically confirmed solid tumor malignancy that is locally advanced or metastatic
6. Disease that is currently refractory to, or not amenable to, standard therapy and/or subjects who are unwilling to try standard chemotherapy
7. Disease that is currently not amenable to surgical intervention, due to either medical contraindications or non-resectability of the tumor
8. Karnofsky performance status ≥ 70%
9. Life expectancy ≥ 3 months, as judged by the investigator
10. No childbearing potential; or use of a medically acceptable form of contraception during the study through the end of follow-up period

Exclusion Criteria:

1. Pregnant or lactating women
2. Primary CNS malignancy and/or active CNS metastases (or leptomeningeal disease) not controlled by prior surgery or radiotherapy
3. Hematologic malignancies (including leukemia of any form, lymphoma, and multiple myeloma)
4. Active second malignancy or history of another malignancy within 2 years with the exception of:

   * Treated, non-melanoma skin cancers
   * Treated carcinoma in situ (CIS) of the breast or cervix
   * Controlled, superficial carcinoma of the bladder
   * T1a or b prostate carcinoma comprising < 5% of resected tissue, with prostate specific antigen (PSA) within normal limits (WNL) since resection
5. Any of the following hematologic abnormalities:

   * Hemoglobin ≤ 9.0 g/dL
   * ANC ≤ 1500 per mm3
   * Platelet count ≤ 75,000 per mm3
6. Any of the following serum chemistry abnormalities:

   * Total bilirubin > 1.5 × the ULN
   * AST or ALT ≥ 3 × ULN (≥ 5 × ULN if due to hepatic involvement by tumor)
   * Serum albumin < 2.5 g/dL
   * Creatinine ≥ 1.5 × ULN
7. Significant cardiovascular disease or condition, including:

   * Congestive heart failure requiring therapy
   * Ventricular arrhythmia requiring therapy
   * Severe conduction disturbance (including QTc interval prolongation > 0.47 sec [corrected], history of a severe arrhythmia, or history of a familial arrhythmia [eg, Wolff-Parkinson-White syndrome])
   * Angina pectoris requiring therapy
   * Left ventricular ejection fraction (LVEF) < 50% by MUGA or echocardiogram
   * Uncontrolled hypertension (as determined by investigator)
   * Myocardial infarction (MI) within 6 months prior to administration of first dose
   * >Class I cardiovascular disease according to the New York Heart Association's (NYHA) Functional Criteria
8. Significant gastrointestinal abnormalities, including:

   * Requirement for IV alimentation
   * Prior surgical procedures affecting absorption
   * Active peptic ulcer disease

     * Grade 2 diarrhea due to any etiology
   * Ulcerative colitis or Crohn's disease
9. Known history of significant ophthalmologic abnormalities, including:

   * Severe dry eye syndrome
   * Keratoconjunctivitis sicca
   * Sjogren's syndrome
   * Severe exposure keratopathy
   * Disorders that might increase the risk for epithelium-related complications (eg, bullous keratopathy, aniridia, severe chemical burns, neutrophilic keratitis)
10. Serious/active infection or any infection requiring parenteral antibiotics
11. Inadequate recovery from prior antineoplastic therapy
12. Inadequate recovery from any prior surgical procedure or major surgical procedure within 2 weeks prior to administration of first dose
13. Life-threatening illness, or organ system dysfunction which, in the opinion of the investigator, would limit life expectancy to < 3 months, compromise the subject's safety, or interfere with evaluation of the safety of the study drug
14. Psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study procedures
15. Inability to comply with the protocol requirements

Drugs and Treatments to be Excluded:

1. Any prior therapy with the following:

   * Doxorubicin at a cumulative dose > 450 mg/m2 or equivalent dose of another anthracycline (eg, daunorubicin, epirubicin, idarubicin) or anthracenedione (eg, mitoxantrone).
   * HKI-272 or any other irreversible EGFR tyrosine kinase inhibitor (eg, CI- 1033 and similar agents).
2. Therapy within 2 weeks prior to administration of the first dose or at any time during the study with:

   • Herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components)
3. Therapy within 3 weeks prior to administration of the first dose or at any time during the study with:

   * Erlotinib (Tarceva®) or gefitinib (Iressa®)
   * Antibodies to EGFR (eg, cetuximab, panitumumab)
   * Agents targeting HER2 (ErbB2) (eg, trastuzumab, lapatinib)
4. Therapy within 4 weeks prior to administration of the first dose or at any time during the study with:

   * Chemotherapy with the exception of the following:
   * Mitomycin C or nitrosoureas within 6 weeks prior to administration of first dose
   * High-dose chemotherapy with stem cell support within 6 months prior to administration of first dose
   * Other antineoplastic agents (standard or therapeutic) for primary malignancy, including but not limited to signal transduction inhibitors and monoclonal antibodies.
   * Immunotherapy, cancer vaccines, biological response modifiers
5. Systemic hormonal therapy within 4 weeks prior to administration of the first dose or at any time during the study, with the exception of the following allowed therapies:

   * Hormonal therapy for appetite stimulation or contraception
   * Nasal, ophthalmic, and topical glucocorticoid preparations
   * Oral replacement therapy for adrenal insufficiency
   * Stable hormonal therapy for prostate carcinoma
   * Low-dose maintenance, or short course (ie, 7 days) steroid therapy for other conditions
6. Any experimental therapy within 4 weeks prior to or at any time during the study
7. Radiotherapy for the primary malignancy:

   * Within 2 weeks prior to first study drug administration if involving ≤25% of marrow-containing bone
   * Within 4 weeks prior to first study drug administration if involving >25% of marrow-containing bone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability, dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of AV-412 administered orally 3 times weekly and once weekly in subjects with relapsed or refractory solid tumor malignancies. | 4 weeks (1 cycle)

SECONDARY OUTCOMES:
Characterize the pharmacokinetic (PK) profile of AV-412 | 8 weeks ( 2 cycles)
Determine the effect of AV-412 on global and targeted gene expression patterns in blood from all subjects enrolled in the MTD expansion cohorts | 8 weeks (2 cycles)
Evaluate the antineoplastic activity of AV-412 | 8 weeks (2 cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Bhargava, M.D., Study Director — AVEO Pharmaceuticals
Locations (4):
- United States (4):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Kansas Masonic Cancer Research Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Montefiore Medical Center, New York, New York